CLINICAL TRIAL: NCT03077035
Title: Using ICDAS II and KaVo DIAGNOdent Pen Detecting Tooth Pit and Fissure Level Incipent Caries Progression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheng-Chao Wang (Other)
Responsible Party: Sponsor-Investigator, Sheng-Chao Wang, Director, Preventive Dentistry Department, Clinical Professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GJ-02
Record Dates: First submitted 2017-02-23; First posted 2017-03-10 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Dental Caries on Pit and Fissure Surface
Keywords: ICDAS; DIAGNOdent; glass ionomer sealant; resin-based sealant; pit and fissure sealants; effectiveness of preventing caries
MeSH Terms: conditions — Van der Woude syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- glass ionomer sealant (Experimental)
  Interventions: Other: glass ionomer sealants
- resin-based sealant (Active Comparator)
  Interventions: Other: resin-based sealant

INTERVENTIONS:
Other: glass ionomer sealants
  Arms: glass ionomer sealant
Other: resin-based sealant
  Arms: resin-based sealant

SUMMARY:
The study was to monitor effectiveness of glass ionomer sealant and resin-based sealant in ICDAS, and to evaluat the correlation between ICDAS and DIAGNOdent over 24 months. Over 200 8-year-old children with at least 2 permanent molar with the International Caries Detection and Assessment System (ICDAS) scores 0-4 were placed glass ionomer sealant and resin-based sealant split-mouthed randomly, and examined with ICDAS and DIAGNOdent before sealents placement and 6, 12 and 24 months after.

ELIGIBILITY:
Inclusion Criteria:

* Subjects provided written informed consent;
* They were 7 to 9 years old;
* They have at least 2 permanent molar with the International Caries Detection and Assessment System (ICDAS) scores 0-4;
* They were generally heallthy

Exclusion Criteria:

* They were allergic to the constituents in pit and fissure sealants

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-10-01 (Estimated); Study Completion 2017-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Decayed Surfaces (DS) of Different Fissure Sealants | Baseline, 6 months, 12 months and 24 months
  Count of DS in different ICDAS cut-off( including D1-6S, D1-2S, D3-6S, D4-6S and D5-6S) in the baseline and 6-month, 12-month and 24-month follow-up.
Change in Repaired Sealants by the baseline ICDAS | 6 months, 12 months and 24 months
  Evaluation the numbers of tooth surface in which the fissure sealants were in the status partially retained or completely lost, and ICDAS score were increasing from the baseline to the 3 follow-ups.
Change in DIAGNOdent Score | Baseline, 6 months, 12 months and 24 months
  The peak value of DIAGNOdent was recorded after repeating it 3 times in the baseline and 3 follow-ups

CONTACTS AND LOCATIONS:
Locations (1):
- School of Stomatology The Fourth Military Medical University, Xi'an, Shaanxi, China